CLINICAL TRIAL: NCT01079052
Title: A Relative Bioavailability Study of 20 mg Famotidine Tablets Under Fed Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 263_FAMOT_07
Record Dates: First submitted 2010-02-18; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Famotidine tablets fed study
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Famotidine Tablets, USP 20 mg of OHM Laboratories Inc (A subsidiary of Ranbaxy Pharmaceuticals Inc., USA)
  Interventions: Drug: Famotidine
- Reference (Active Comparator): Pepcid® AC Acid reducer famotidine tablets 20 mg of Johnson & Johnson. Merck Consumer Pharmaceutical Co. Fort Washington, PA 19034 USA
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Famotidine — Tablets

SUMMARY:
The study was conducted as an open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioavailability study comparing famotidine tablets, USP 20 mg manufactured by OHM Laboratories with Pepcid® AC Acid reducer famotidine tablets 20 mg (containing famotidine 20 mg) distributed by Johnson & Johnson. Merck Consumer Pharmaceutical Co. Fort Washington, PA 19034 USA under fed conditions.

DETAILED DESCRIPTION:
Following an overnight fast of at least 10 hours, all subjects were served a high-fat high-calorie breakfast. Thirty minutes after the start of the breakfast, subjects were administered a single oral dose of famotidine tablets, USP 20 mg or Pepcid® AC Acid reducer famotidine tablets 20 mg (containing famotidine 20 mg) under low-light condition during each period of the study, along with 240 mL of drinking water at ambient temperature and under supervision of trained study personnel.

During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis) at baseline. Adverse event monitoring was done throughout the study. Laboratory parameters of hematology and biochemistry (except blood glucose and cholesterol) were repeated at the end of the study for all the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for their corresponding height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.
* Had a non-vegetarian diet habit.

There were no deviations in this regard.

Exclusion Criteria:

* History of hypersensitivity to famotidine and/or related group of drugs, including hypersensitivity to other H2 blockers.
* The subject had evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Presence of values which were significantly different from normal reference range and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
* Presence of values which were significantly different from normal reference range and/or judged clinically significant for serum creatinine, blood urea, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray.
* The subject had history of serious gastrointestinal, hepatic, renal, pulmonary, cardiovascular, neurological or haematological disease, diabetes or glaucoma.
* The subject had history of any psychiatric illness, which might impair the ability to provide written informed consent.
* The subject was a regular smoker who smoked more than 10 cigarettes daily or has difficulty abstaining from smoking for the duration of each study period.
* The subject had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* The subject had participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

There were no deviations in this regard.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of ranbaxy famotidine tablets 20mg with Pepcid® AC Acid reducer famotidine tablets 20 mg under fed condition

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Clinical Pharmacology Unit, Ranbaxy Laboratories Limited, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html